CLINICAL TRIAL: NCT03251846
Title: Pediatrics Owning Performance Study
Acronym: POPS!
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Children's Hospitals and Clinics of Minnesota (Other)
Collaborators: Pops! Diabetes Care (Unknown)
Responsible Party: Principal Investigator, Laura Gandrud, Principal Investigator, Children's Hospitals and Clinics of Minnesota
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1704-059
Record Dates: First submitted 2017-08-14; First posted 2017-08-16 (Actual); Last update posted 2017-08-17 (Actual); Status verified 2017-08

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Diabetes Mellitus, Type 1; self-monitoring blood glucose; diabetes mobile application; diabetes management device
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: prospective, single-arm, single-subject clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

INTERVENTIONS:
Device: Pops! One personalized mobile platform — Enrolled subjects will be given a POPS! Device (meter, lancet/test strips, and software app) to use for 6 months. Primary outcomes will be measured at baseline and 6-month follow-up.

SUMMARY:
A more convenient blood glucose monitoring system integrated with a responsive mobile health app may facilitate improved diabetes control in adolescent and young adult patients with Type 1 diabetes. The primary aim of this study is to determine if the POPS diabetes management system can improve diabetes control in the adolescent and young adult population. The investigators hypothesize that use of the POPS diabetes management device and mobile application (app) will be associated with lower HbA1C after 6-months of use in adolescent and young adult T1D patients.

DETAILED DESCRIPTION:
This is a prospective, single-arm, single-subject clinical trial to study outcomes related to device use in the pediatric diabetes population. Patients will be recruited at the Children's Minnesota McNeely Diabetes Clinic and satellite clinics during routine office visits over a 6-month period until recruitment goals are met. Enrolled subjects will be given a POPS! Device (meter, lancet/test strips, and software app) to use for 6 months with periodic check-ins and follow-ups. Primary outcome, HbA1c, will be measured at baseline and 6-month follow-up. Secondary aims include assessment of blood glucose testing frequency and quality of life scores following 6-months of device and app use. The investigators will also describe sustained use over the study period, average blood glucose and variability, and frequency of hypoglycemic events (blood glucose <70). Historical data for each patient will also be recorded from medical records, with each patient serving as their own comparative control.

ELIGIBILITY:
Inclusion Criteria:

1. Type 1 diabetes, diagnosed at least 6 months prior to enrollment
2. Aged ≥10 years, ≤25 years
3. Daily insulin of any type, administered as multiple daily injections (MDI) for at least 90 days prior to enrollment
4. Latest HbA1c ≥8.0%, ≤10.5%
5. Average self-blood glucose measurement frequency ≥2 per day and ≤4.5 per day based on meter download spanning 28-day period prior to qualifying HbA1c measurement
6. User of iPhone 5 or above with iOS above 10.0
7. English-speaking
8. Patient must be willing to only use POPS device to check blood glucose for duration of study (except in case of technical failure or emergency)

Exclusion Criteria:

1. Continuous glucose monitor user at time of enrollment or considering CGM use in the next 6 months
2. Concurrent participation in another study that may influence results
3. On insulin pump at time of recruitment or considering pump use in the next 6 months
4. Inability to perform self-care behaviors due to co-morbidities such as mental health disorder, developmental delay, or other prohibitive physical condition (blindness, etc)
5. Participation in a diabetes clinical trial intervention in the 12 months prior to enrollment

Ages: 10 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-07-17 (Actual); Primary Completion 2018-07 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
HbA1c | 6 months
  Change in HbA1c from baseline to 6 months

SECONDARY OUTCOMES:
Testing frequency | 30 days prior to enrollment to 6 months post-enrollment
  Blood glucose testing frequency
quality of life | 30 days prior to enrollment to 6 months post-enrollment
  Peds QL diabetes module
Average blood glucose | 30 days prior to enrollment to 6 months post-enrollment
  Average blood glucose during 30 days prior to enrollment and during the 6 month intervention
Blood glucose variability | 30 days prior to enrollment to 6 months post-enrollment
  Blood glucose variability during 30 during prior to enrollment and during the 6 months of intervention
Hypoglycemia | 6 months
  Frequency of hypoglycemic events during intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospitals and Clinics of Minnesota, Saint Paul, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No